CLINICAL TRIAL: NCT04244071
Title: The Effect of Active and Passive Heating Methods Used in Different Areas of Perioperative Processes on Thermal Comfort and Anxiety
Brief Title: The Effect of Heating on Thermal Comfort and Anxiety
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Selcuk University (Other)
Collaborators: Koç University (Other)
Responsible Party: Principal Investigator, Tunc Tuna Pinar, PhD, Research Asistant, Selcuk University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Selcuk
Record Dates: First submitted 2020-01-21; First posted 2020-01-28 (Actual); Last update posted 2020-01-28 (Actual); Status verified 2020-01

CONDITIONS: Anxiety; Nurse-Patient Relations
Keywords: nursing; active heating; thermal comfort; anxiety
MeSH Terms: conditions — Anxiety Disorders | interventions — Patient Health Questionnaire

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- Group C (Active Comparator): Usual care (Group C): The patients in this group received routine hospital care.
  Vital signs, thermal comfort, and anxiety levels of the patients were evaluated.
  Interventions: Other: routine hospital care
- Group A (Experimental): The patients in Group A were warmed up using a gown blowing warm air starting at least 30 min prior to the surgery until they were anesthetized.
  Vital signs, thermal comfort, and anxiety levels of the patients were evaluated.
  Interventions: Device: Bair Paws Blanket 81003 and FOC device 87500
- Group B (Experimental): Routine care was provided for the patients in Group B in the preoperative and intraoperative periods. In the postoperative period, patients were warmed up using a gown blowing warm air after they were transferred to the post-anesthesia care unit, and continued to be warmed up on the basis of the temperature set by themselves until they wore their own clothes in the ward.
  Vital signs, thermal comfort, and anxiety levels of the patients were evaluated.
  Interventions: Device: Bair Paws Blanket 81003 and FOC device 87500; Other: routine hospital care

INTERVENTIONS:
Device: Bair Paws Blanket 81003 and FOC device 87500 — This study is a randomized, pretest - posttest controlled experimental design.
  Other Names: Thermal Comfort Scale; Anxiety Scale
  Arms: Group A; Group B
Other: routine hospital care — routine hospital care
  Arms: Group B; Group C

SUMMARY:
This study with a randomized, pretest - posttest controlled experimental design was conducted to determine the effects of active and passive heating methods applied in different parts of the perioperative process on thermal comfort, anxiety and vital signs. The study was conducted with the patients who were hospitalized for open abdominal surgical interventions in the Department of Obstetrics and Gynecology, of Selcuk University Medical Faculty Hospital, between the dates of 1 October 2018 and 10 January 2019. The study included 99 patients in two control groups and one experimental group. The patients in group A were dressed with hot air blowing patients scrubs in both preoperative and postoperative periods, while patients in group B were dressed with hot air blowing patients scrubs only in the postoperative period. The control group continued routine practice. In the preoperative period, vital signs, thermal comfort, and anxiety levels of the patients were evaluated. In the intraoperative period, vital signs and thermal comfort levels of the patients were evaluated. Thermal comfort level of the patients was re-evaluated prior to the induction of anesthesia. Once the patients were transferred to the post-anesthesia care unit, among the vital signs of the patients, body temperature was measured in the temporal region, and other signs were measured using the monitors. Thermal comfort and anxiety levels of the patients were re-evaluated after they got dressed.

DETAILED DESCRIPTION:
"Perioperative hypothermia," which is defined as a decrease below 36 °C in the body temperature 1 h prior to anesthesia and up to 24 h following anesthesia is a common problem in patients undergoing surgery. Perioperative hypothermia leads to many problems.

Given the negative effects of increased anxiety and deterioration in thermal comfort due to perioperative hypothermia (such as decreased satisfaction and increased pain) hypothermia poses a problem that should be highlighted and prevented. It is also important for nurses to understand hypothermia and the complications associated with it and take effective measures. In the present randomized controlled trials, gowns blowing warm air; heated blankets, fabrics, and liquid; and self-heating blankets were used for increasing thermal comfort. No common heating technique or heating area was used in these studies In this context, the primary purpose of the present study was to determine the effects of active (gown blowing warm air) and passive (heated blanket) heating on thermal comfort and anxiety in preoperative and postoperative periods in patients scheduled for open abdominal surgery.

ELIGIBILITY:
Inclusion Criteria:

* Being scheduled for open abdominal surgery
* Being an inpatient in the obstetrics and gynecology ward
* 2-4 h surgery duration
* 1 and 2 ASA scores
* Being able to speak Turkish
* Being 18-65 years of age

Exclusion Criteria:

* Mental retardation and psychiatric disorder,
* The presence of severe lesions or wounds on the skin
* Being an alcohol and drug addict

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2018-03-30 (Actual); Primary Completion 2019-01-10 (Actual); Study Completion 2019-05-30 (Actual)

PRIMARY OUTCOMES:
Thermal comfort | baseline (at the beginning of treatment)
  Thermal comfort level was measured using a 10-cm visual analog scale, The patients were explained that 1 point indicated "no comfort" and 10 points indicated "the highest level of comfort," and then they were asked to give 1-10 points for their comfort levels.
Anxiety | baseline (at the beginning of treatment)
  The state-trait anxiety inventory developed by Spielberger et al. (1970) was used to measure the anxiety levels of the patients. The state anxiety inventory evaluates "how one feels at a certain moment and under certain conditions," whereas the continuous anxiety inventory evaluates "how one feels irrespective of the circumstances and conditions that he or she is in." A high score is an indicator of high anxiety level

SECONDARY OUTCOMES:
Body temperatures | baseline (at the beginning of treatment)
  In the evaluation of life findings of patients in the perioperative period; ARMOLINE contactless electronic infrared thermometer was used for fire. (degrees centigrade)
blood pressure values | baseline (at the beginning of treatment)
  In the evaluation of life findings of patients in the perioperative period; GAMMA brand sphygmomanometer was used for blood pressure. (mm Hg)
pulse values | baseline (at the beginning of treatment)
  In the evaluation of life findings of patients in the perioperative period; plusMED -50DL finger-type pulse oximeter was used to measure saturation. (beats per minute)
respiratory rates | baseline (at the beginning of treatment)
  the respiratory rate was counted for one minute. (beats per minute)
saturation values | baseline (at the beginning of treatment)
  In the evaluation of life findings of patients in the perioperative period; plusMED -50DL finger-type pulse oximeter was used to measure saturation. (PO2)

CONTACTS AND LOCATIONS:
Overall Officials: Pinar Tunc Tuna, Study Director — Selcuk Universty; Serife Kursun, Study Director — Selcuk Universty; Inci Kara, Study Director — Selcuk Universty
Locations (1):
- Selcuk Universty, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No